CLINICAL TRIAL: NCT02248961
Title: Open-label, Randomized, Multicenter, Efficacy and Safety Evaluating Study to Compare Kanarb (Fimasartan), Manufactured by Boryung Pharmaceutical Co., Ltd, Republic of Korea, Tablets 60/120 mg and Cozaar® (Losartan), Manufactured by MERCK SHARP & DOHME B.V., Netherlands, Tablet 50/100 mg in Adult Patients With Grade I-II Arterial Hypertension
Brief Title: Efficacy and Safety Evaluating Study to Compare Kanarb (Fimasartan) and Cozaar® (Losartan) in Adult Patients With Grade I-II Arterial Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: R-Pharm (Industry)
Collaborators: Covance (Industry); Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC09042014
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-02

CONDITIONS: Arterial Hypertension
MeSH Terms: conditions — Hypertension | interventions — fimasartan; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kanarb (Fimasartan) (Experimental): 88 subjects will receive Kanarb (Fimasartan), manufactured by Boryung Pharmaceutical Co., Ltd, Republic of Korea, tablets 60/120 mg for 12 weeks
  Interventions: Drug: Fimasartan
- Cozaar® (Losartan) (Active Comparator): 88 subjects will receive Cozaar® (Losartan), manufactured by MERCK SHARP & DOHME B.V., Netherlands, tablets 50/100 mg for 12 weeks
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Fimasartan — Starting dose of Kanarb (Fimasartan) is 60 mg, orally, once a day in the morning. The subjects will visit the clinical site every 4 weeks to measure Arterial blood pressure (ABP). The dose will be doubled in case if SBP ≥140 mmHg or DBP ≥90 mmHg at Visit 3 (Day 28) or at Visit 4 (Day 56).
  If necessary, the dose of the study drug may be increased based on the assessment of patient's condition performed at the phone contact (Day14±3). Patient may be called for an unscheduled visit for treatment adjustment (decided individually, with possibility of dose titration as per investigator's judgment, indicated in source documents).
  When possibilities are, the patient should be administrated by the study medication at the same time in the morning.
  Other Names: Kanarb
  Arms: Kanarb (Fimasartan)
Drug: Losartan — Cozaar® (Losartan), manufactured by MERCK SHARP & DOHME B.V., Netherlands, tablets 50/100 mg
  Other Names: Cozaar®
  Arms: Cozaar® (Losartan)

SUMMARY:
Assess and compare the efficacy and safety of Kanarb (Fimasartan), manufactured by Boryung Pharmaceutical Co., Ltd, Republic of Korea, tablets 60/120 mg and Cozaar® (Losartan), manufactured by MERCK SHARP & DOHME B.V., Netherlands, tablet 50/100 mg in adult patients with Grade I-II arterial hypertension in 12 weeks of therapy

DETAILED DESCRIPTION:
1. To evaluate efficacy of 12-week Kanarb (Fimasartan), manufactured by Boryung Pharmaceutical Co., Ltd, Republic of Korea, tablets 60/120 mg and Cozaar® (Losartan), manufactured by MERCK SHARP & DOHME B.V., Netherlands, tablet 50/100 mg in adult patients with Grade I-II arterial hypertension.
2. To evaluate safety of 12-week Kanarb (Fimasartan), manufactured by Boryung Pharmaceutical Co., Ltd, Republic of Korea, tablets 60/120 mg and Cozaar® (Losartan), manufactured by MERCK SHARP & DOHME B.V., Netherlands, tablet 50/100 mg in adult patients with Grade I-II arterial hypertension.
3. Assess the pharmacokinetics parameters of Kanarb (Fimasartan), manufactured by Boryung Pharmaceutical Co., Ltd, Republic of Korea in adult patients with arterial hypertension I-II stage after a single dose.

Starting dose of Kanarb (Fimasartan), manufactured by Boryung Pharmaceutical Co., Ltd, Republic of Korea is 60 mg, orally, once a day in the morning.

The planned study duration for each subject is 18 weeks maximum:

The screening period could takes up to 2 weeks (including the 1-week "wash-out" period ) - the screening period duration depends on the prior anti-hypertensive therapy:

* "naive" subjects who never received therapy (which must be reflected in the source documents), may be randomized after completion of all screening procedures;
* Subjects receiving anti-hypertensive therapy which may be discontinued without prior dose reduction must undergo a 7 days "wash-out" period, so the screening period will take at least 7 days;
* Subjects, receiving anti-hypertensive therapy which requires dose reduction before discontinuation must undergo the 7 days "wash-out" period after the last dose administration, so the screening period will consist of dose reduction period and a "wash-out" period.

Treatment period - 12 weeks. Follow-up period - 4 weeks. The subjects will visit the clinical site every 4 weeks to measure ABP. The dose will be doubled in case if SBP ≥140 mmHg or DBP ≥90 mmHg at Visit 3 (Day 28) or at Visit 4 (Day 56).

If necessary, the dose of the study drug may be increased based on the assessment of patient's condition performed at the phone contact (Day14±3). Patient may be called for an unscheduled visit for treatment adjustment (decided individually, with possibility of dose titration as per investigator's judgment, indicated in source documents).

When possibilities are, the patient should be administrated by the study medication at the same time in the morning. Governing conditions for defining the time of the drug administration is the subject comfort and the time of its visits the research center.

If laboratory tests are scheduled, a patient should come to the research center fasting (food is prohibited for 8 hours before the visit).

All of the clinical evaluations are conducted on the next morning after taking the medication. On the visit day a patient comes to the research center not taking the drug, and after all the planned procedures are conducted the patient is administrated by the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of both sex aged 18-75 inclusively.
2. Subjects who signed their written Informed Consent for participation in the study and willing to adhere to all Protocol procedures.
3. Subjects with documented diagnosis of grade I-II primary arterial hypertension within at least 3 months before screening.
4. Systolic blood pressure (SBP) (when seated) at Screening (Day -14)

   * For subjects administered with anti-hypertensive therapy: SBP ≤ 179 Hg
   * For subjects receiving no anti-hypertensive therapy (so called 'naïve' patients): 140≥SBP ≤179.
5. As per investigator's judgment, subjects with controlled arterial hypertension must benefit from the therapy switch to Kanarb (Fimasartan), manufactured by Boryung Pharmaceutical Co., Ltd, Republic of Korea, tablets 60/120 mg and Cozaar® (Losartan), manufactured by MERCK SHARP & DOHME B.V., Netherlands, .
6. For subjects administered with anti-hypertensive drugs: the anti-hypertensive drug may be safely cancelled during the "wash-out" period according to the investigator's judgment.
7. For women of child-bearing potential: negative urine pregnancy test at screening (Day -14). 8. Systolic blood pressure (SBP) (when seated) at Randomization (Day 0) ≥140 mmHg and ≤179 mmHg.

9. For women of child-bearing potential: negative urine pregnancy test at Randomization (Day 0)

Exclusion Criteria:

1. Grade III Arterial Hypertension.
2. Arterial hypotension (SPB ≤100 mm Hg) at Screening (Day -14) and/or Randomization (Day 0).
3. Subjects needing treatment with more than one anti-hypertensive drug (more than one active substance, including complex drugs).
4. Secondary (symptomatic) arterial hypertension.
5. Known bilateral renal arterial stenosis or unilateral renal arterial stenosis.
6. Hyperpotassemia >5,0 mmol/l (as per blood biochemistry results at Screening).
7. Primary hyperaldosteronism.
8. Known hypersensitivity to angiotensin-II receptors antagonists or any other study drug or comparator component.
9. Contraindications for use of angiotensin-II receptors antagonists.
10. Myocardial infarction and or unstable angina, and/or acute cerebrovascular accident/transient ischemic attack, and/or percutaneous coronary intervention, and/or coronary arterial bypass graft, acute coronary arteries involvement, and/or obliterative vascular atherosclerosis of low extremities, and/or grade III and IV retinopathy in anamnesis.
11. Clinically significant cardiac valves damage.
12. Cardiomyopathies
13. Chronic Heart failure (CHF) (except for CHF FC I NYHA).
14. Creatinine clearance less than 60 ml/min/1.73m2 calculated by Cockroft-Gault formula.
15. Known moderate to severe hepatic insufficiency and/or transaminase increase: AST and/or ALT ≥2*ULN.
16. History of infections (HIV, hepatitis B or C, syphilis).
17. Uncontrolled Diabetes mellitus, Glycosylated hemoglobin level (HbA1c) >7%.
18. Severe systemic diseases, such as gastro-intestinal tract diseases, autoimmune disorders, blood disorders and other conditions which may affect on the study drugs' absorption, distribution and and excretion.
19. Clinically significant abnormalities of laboratory parameters.
20. Drug or alcohol addiction, psychiatric disorders.
21. Medical history of oncological disease within 5 years before screening.
22. Subjects with biliary tracts obstruction.
23. Subjects with genetic disorders, such as galactose intolerance, congenital lactase insufficiency and glucose-galaclose malabsorption syndrome.
24. Any other acute disease or progression and/or decompensation at the moment of enrollment
25. Necessity to administer or administration of prohibited concomitant drugs from the "List of Prohibited Drugs" within 14 days before enrollment
26. Pregnancy or breast-feeding period; fertile women not using adequate contraception methods
27. Participation in another clinical trial within 3 months before Screening.
28. Other medical or psychiatric conditions or lab abnormalities that may increase potential risk associated with study participation and IP administration, or that may affect study results interpretation and as per investigator's judgment, make the subject ineligible.
29. Study site personnel or Sponsor's representatives immediately involved in the study.
30. Subjects, excluded from the study may not be included in it again.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Russia (13):
  - Federal State Institution "Russian Cardiology Research and Production Complex" of the Ministry of Health and Social Development of the Russian Federation (FSI "Cardiology" Russian Healthcare Ministry), Moscow
  - Moscow Health Department "City Clinical Hospital № 81", Moscow
  - State Research Center for Preventive Medicine of Ministry of Health of the Russian gederation, Moscow
  - St. Petersburg State health agency "City Hospital number 38 it. NA Semashko ", Pushkin
  - St. Petersburg State healthcare Institution "City Hospital number 28" "Maximilianovskaya", Saint Petersburg
  - Clinical Hospital n. a. St. Luka, Saint Petersburg
  - Federal Almazov Medical Research Centre, Saint Petersburg
  - St. Petersburg State Healthcare Institution 'Diagnostic Centre #85', Saint Petersburg
  - St. Petersburg State Institution of Health "City Hospital № 15", Saint Petersburg
  - St. Petersburg State Institution of Healthcare "Pokrovskaya City Hospital", Saint Petersburg
  - State Budget Education Institution of Higher Professional Education "North-Western State Medical University named after I.I. Mechnikov" on base St. Petersburg State Institution of Healthcare "Pokrovskaya City Hospital", Saint Petersburg
  - State Budget Education Institution of Higher Professional Education "North-Western State Medical University named after I.I. Mechnikov", the department faculty and hospital care, court number 5, Saint Petersburg
  - Troitsk City Hospital, Troitsk

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruitment was conducted in 13 clinical sites of Moscow and Saint-Petersburg between May and October of 2014
Pre-assignment Details: Duration of screening period was up to 14 days depended on prior antihypertensive treatment. 184 patients were screened, 179 randomized.
Groups:
- Kanarb (Fimasartan): 60/120 mg Kanarb (Fimasartan) administered orally once a day in the morning for 12 weeks period
- Cozaar® (Losartan): 50/100 mg Cozaar® (Losartan) administered orally once a day for 12 week period
Period: Overall Study
Arm/Group | Kanarb (Fimasartan) | Cozaar® (Losartan)
Started | 89 | 90
Completed | 86 | 88
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Unmet inclusion/exclusion criteria | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set Population (FAS) - those subjects from Intent-to-treat population (ITT, all randomized patients), who had at least one assessment for efficacy analysis after the start of therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Kanarb (Fimasartan) | Cozaar® (Losartan) | Total
Number analyzed (Participants) | 89 | 90 | 179
Age, Continuous [Mean (Full Range); unit: years] | 53.4 [25.6 to 75.9] | 53.8 [21.9 to 73.2] | 53.6 [21.9 to 75.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 34 | 64
  Male | 59 | 56 | 115
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  European | 87 | 90 | 177
  Asian | 2 | 0 | 2
BMI [Mean (Full Range); unit: kg/m^2] — Body Mass Index calculated as weight(kg)/height(m^2)
  kg/m^2 | 29.4 [20.3 to 50.5] | 28.9 [20.7 to 41.7] | 29.1 [20.3 to 50.5]
Arterial hypertension (AH) duration [Mean (Full Range); unit: years] — The duration of AH in patients at study inclusion in population of all randomized patients
  years | 5.8 [0.3 to 19.2] | 6.2 [0.3 to 33.1] | 6.0 [0.3 to 33.1]
Hypertension grade [Count of Participants; unit: Participants] — The grade of blood pressure increase was determined in accordance with Russian guidelines (fourth revision) "Diagnosis and treatment of arterial hypertension".
  Grade I AH: sistolic blood pressure (SBP) 140-159 mmHg and/or diastolic blood pressure (DBP) 90-99 mmHg
  Grade II AH: sistolic blood pressure (SBP) 160-179 mmHg and/or diastolic blood pressure (DBP) 100-109 mmHg
  Participants
    Grade I | 20 | 27 | 47
    Grade II | 69 | 63 | 132
Chronic heart failure (CHF) NYHA Class I [Count of Participants; unit: Participants] — Patients with no limitation of physical activity (ordinary physical activity does not cause undue fatigue, palpitation, dyspnea - shortness of breath) but having symptoms of chronic heart failure could be defined as NYHA (New-York Heart Association) Class I of chronic heart failure
  Participants | 10 | 12 | 22
Prior therapy for arterial hypertension [Count of Participants; unit: Participants] | 55 | 46 | 101
Smoking history [Count of Participants; unit: Participants]
  Smoker | 19 | 62 | 81
  Has never smoked | 63 | 21 | 84
  Smoker-in-the-past | 7 | 7 | 14
Alcohol history [Count of Participants; unit: Participants]
  Drinking | 52 | 57 | 109
  Never-drinking | 25 | 23 | 48
  Drinking-in-the-past | 12 | 9 | 21
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure (SBP) After 12 Weeks of Treatment
Description: The value of SBP (seated) to be registered was mean of the 3 measurements performed with interval no less than 1 minute using the manual (mercury or mechanic) tonometer after 5 minutes rest.
  "Change" was calculated as (Value of SBP at week 12 minus Value of SBP at baseline).
Time Frame: Baseline and week 12 of treatment
Population: Full Analysis Set Population (FAS) - those subjects from Intent-to-treat population (ITT, all randomized patients), who had at least one assessment for efficacy analysis after the start of therapy. Last observation carried forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Kanarb (Fimasartan) | Cozaar® (Losartan)
Number analyzed (Participants) | 89 | 90
mm Hg
  SBP at Baseline | 152.9 (5.9) | 151.9 (5.9)
  Change from Baseline at Week 12 | -25.2 (8.6) | -24.3 (7.8)
Statistical Analysis 1: Comparison: Kanarb (Fimasartan) vs Cozaar® (Losartan); The null hypothesis (H0) is that there is a decrease in SBP on the background treatment with Kanarb (fimasartan), that is at least 5.5 mmHg lower compared to Cozaar® (losartan). Test of the hypotheses was performed using mixed linear models, where the site effect was considered a random effect, and the treatment group effect was considered a fixed effect. Baseline SBP on the study arm was included into the model as a covariate (a fixed effect) in all cases; Test type: Other — It was calculated that at least 140 patients (70 patients per group) must be enrolled into the study to achieve 80% power. With regard to 20% of patients withdrawn prematurely or data not suitable for analysis, it was necessary to include at least 176 patients (88 per group) into the study; p = 0.390, Mixed Models Analysis; Mean Difference (Final Values) = -0.18, 95% CI 1-sided [upper limit 1.47], Standard Error of Mean 1.00

2. Secondary Outcome: Change in Diastolic Blood Pressure (DBP) After 4 Weeks of Treatment
Description: The value of DBP (seated) to be registered was mean of the 3 measurements performed with interval no less than 1 minute using the manual (mercury or mechanic) tonometer after 5 minutes rest.
  "Change" was calculated as (Value of DBP at week 4 minus Value of SBP at baseline).
Time Frame: Baseline and week 4 of treatment
Population: All randomized patients, who had at least one assessment for efficacy analysis after the start of therapy. One patient (Kanarb (fimasartan) treatment group) was withdrawn from the study by the time of assessment at week 4.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Kanarb (Fimasartan) | Cozaar® (Losartan)
Number analyzed (Participants) | 89 | 90
mm Hg
  DBP at Baseline | 88.7 (8.1) | 89.6 (6.9)
  Change from Baseline at Week 4: number analyzed (Participants) | 88 | 90
  Change from Baseline at Week 4 | -9.5 (9.1) | -7.4 (7.5)
Statistical Analysis 1: Comparison: Kanarb (Fimasartan) vs Cozaar® (Losartan); Test type: Other; p = 0.018, Mixed Models Analysis; The investigational site was included as random effect. The baseline levels of SBP and the treatment group were included as fixed effects

3. Secondary Outcome: Change in DBP After 8 Weeks of Treatment
Description: The value of DBP (seated) to be registered was mean of the 3 measurements performed with interval no less than 1 minute using the manual (mercury or mechanic) tonometer after 5 minutes rest.
  "Change" was calculated as (Value of DBP at week 8 minus Value of SBP at baseline).
Time Frame: Baseline and week 8 of treatment
Population: All randomized patients, who had at least one assessment for efficacy analysis after the start of therapy. One patient (Kanarb (fimasartan) treatment group) was withdrawn from the study by the time of assessment at week 8.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Kanarb (Fimasartan) | Cozaar® (Losartan)
Number analyzed (Participants) | 89 | 90
mm Hg
  DBP at Baseline | 88.7 (8.1) | 89.6 (6.9)
  Change from Baseline at Week 8: number analyzed (Participants) | 88 | 90
  Change from Baseline at Week 8 | -10.3 (9.5) | -10.7 (7.9)
Statistical Analysis 1: Comparison: Kanarb (Fimasartan) vs Cozaar® (Losartan); Test type: Other; p = 0.579, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: Change in DBP After 12 Weeks of Treatment
Description: The value of DBP (seated) to be registered was mean of the 3 measurements performed with interval no less than 1 minute using the manual (mercury or mechanic) tonometer after 5 minutes rest.
  "Change" was calculated as (Value of DBP at week 12 minus Value of SBP at baseline).
Time Frame: Baseline and week 12 of treatment
Population: One patient (Kanarb (fimasartan) treatment group) was withdrawn from the study by the time of assessment at week 12
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Kanarb (Fimasartan) | Cozaar® (Losartan)
Number analyzed (Participants) | 89 | 88
mm Hg
  DBP at Baseline | 88.7 (8.1) | 89.6 (6.9)
  Change from Baseline at Week 12: number analyzed (Participants) | 88 | 88
  Change from Baseline at Week 12 | -10.6 (8.8) | -11.3 (7.8)
Statistical Analysis 1: Comparison: Kanarb (Fimasartan) vs Cozaar® (Losartan); Test type: Other; p = 0.466, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

5. Secondary Outcome: Change in SBP After 4 Weeks of Treatment
Description: The value of SBP (seated) to be registered was mean of the 3 measurements performed with interval no less than 1 minute using the manual (mercury or mechanic) tonometer after 5 minutes rest.
  "Change" was calculated as (Value of SBP at week 4 minus Value of SBP at baseline).
Time Frame: Baseline and week 4 of treatment
Population: One patient (Kanarb (fimasartan) treatment group) was withdrawn from the study by the time of assessment at week 4
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Kanarb (Fimasartan) | Cozaar® (Losartan)
Number analyzed (Participants) | 89 | 90
mm Hg
  SBP at Baseline | 152.9 (5.9) | 151.9 (5.9)
  Change from Baseline at Week 4: number analyzed (Participants) | 88 | 90
  Change from Baseline at Week 4 | -19.7 (10.3) | -17.6 (10.5)
Statistical Analysis 1: Comparison: Kanarb (Fimasartan) vs Cozaar® (Losartan); Test type: Other; p = 0.118, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

6. Secondary Outcome: Change in SBP After 8 Weeks of Treatment
Description: The value of SBP( seated) to be registered was mean of the 3 measurements performed with interval no less than 1 minute using the manual (mercury or mechanic) tonometer after 5 minutes rest.
  "Change" was calculated as (Value of SBP at week 8 minus Value of SBP at baseline).
Time Frame: Baseline and week 8 of treatment
Population: One patient (Kanarb (fimasartan) treatment group) was withdrawn from the study by the time of assessment at week 8
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Kanarb (Fimasartan) | Cozaar® (Losartan)
Number analyzed (Participants) | 89 | 90
mm Hg
  SBP at Baseline | 152.9 (5.9) | 151.9 (5.9)
  Change from Baseline at Week 8 | -23.5 (9.0) | -23.9 (8.6)
Statistical Analysis 1: Comparison: Kanarb (Fimasartan) vs Cozaar® (Losartan); Test type: Other; p = 0.662, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

7. Secondary Outcome: Number of Subjects Who Responded on Therapy
Description: The subject will be considered a responder if SBP (when seated) <140 mmHg or SBP decrease is >10% from baseline.
Time Frame: Week 12 of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Kanarb (Fimasartan) | Cozaar® (Losartan)
Number analyzed (Participants) | 89 | 90
Participants | 85 | 90
Statistical Analysis 1: Comparison: Kanarb (Fimasartan) vs Cozaar® (Losartan); Test type: Other; p = 0.143, Mantel Haenszel

ADVERSE EVENTS:
Time Frame: 18 weeks
Description: The number and percent of subjects and number and group of AEs will be performed within every organ/system group
Arm/Group | Kanarb (Fimasartan) | Cozaar® (Losartan)
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/90
Other Adverse Events (participants affected / at risk) | 20/89 | 15/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Kanarb (Fimasartan) (N=89) | Cozaar® (Losartan) (N=90)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Conjunctival oedema (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Diarrhoea (General disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Bronchitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2
Pharyngitis (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Blood pressure increased (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 0
Low density lipoprotein increased (Investigations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 4 | 3
Renal impairment (Renal and urinary disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study related information could be made public availiable only after Sponsors written permission.